CLINICAL TRIAL: NCT04086745
Title: A Randomized, Controlled Pragmatic Phase 3b/4 Study of Baricitinib in Patients With Rheumatoid Arthritis
Brief Title: A Study of Baricitinib in Participants With Rheumatoid Arthritis
Acronym: RA-BRANCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17363; I4V-MC-JAJD (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — baricitinib; Tumor Necrosis Factor Inhibitors; Etanercept; Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Baricitinib Low Dose (Experimental): Baricitinib administered orally.
  Interventions: Drug: Baricitinib
- Baricitinib High Dose (Experimental): Baricitinib administered orally.
  Interventions: Drug: Baricitinib
- TNF Inhibitor (Active Comparator): Adalimumab or etanercept administered subcutaneously (SC) per standard of care.
  Interventions: Drug: TNF Inhibitor

INTERVENTIONS:
Drug: Baricitinib — Administered orally.
  Other Names: LY3009104
  Arms: Baricitinib High Dose; Baricitinib Low Dose
Drug: TNF Inhibitor — Administered SC
  Other Names: Etanercept; Adalimumab
  Arms: TNF Inhibitor

SUMMARY:
This post-marketing study is designed to compare the safety of baricitinib versus tumor necrosis factor (TNF) inhibitors with respect to venous thromboembolic events (VTEs) when given to participants with rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have at least one of the following characteristics:

  * Documented evidence of a VTE prior to this study
  * At least 60 years of age
  * A body mass index (BMI) greater than or equal to 30 kilograms per meter squared (kg/m²), or
  * Age 50 to less than 60 years and BMI 25 to less than 30 kg/m²
* Participants must have an inadequate response or intolerance to at least 1 disease-modifying antirheumatic drugs (DMARD) (synthetic or biologic)

Exclusion Criteria:

* Participant must not have prior use of a Janus kinase (JAK) inhibitor or have received more than 1 prior TNF inhibitor that was:

  * discontinued for IR (lack or loss of efficacy) for RA, or
  * discontinued for intolerance (AE) when used for any indication
* Participants must not be pregnant or breastfeeding
* Participants must not have had more than one VTE
* Participants must not have cancer
* Participants must not have active herpes zoster, serious infection, active tuberculosis, or any other serious illness
* Participants must not have had a live vaccine within four weeks of study start
* Participants must not have participated in any other clinical trial within four weeks of study start
* Participants must not have a history of IV drug use, other illicit drug abuse, or chronic alcohol abuse in the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1317 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
Time from First Dose of Study Treatment to First Event of Venous Thromboembolism (VTE) | Baseline through Study Completion (Approximately 5.5 Years)
  Time from First Dose of Study Treatment to First Event of VTE

SECONDARY OUTCOMES:
Time from First Dose of Study Treatment to First Arterial Thromboembolic Event (ATE) | Baseline through Study Completion (Approximately 5.5 Years)
  Time from First Dose of Study Treatment to First ATE
Time from First Dose of Study Treatment to First Major Adverse Cerebro-Cardiovascular Event (MACE) | Baseline through Study Completion (Approximately 5.5 Years)
  Time from First Dose of Study Treatment to First MACE
Time from First Dose of Study Treatment to First Malignancy (excluding nonmelanoma skin cancer [NMSC]) | Baseline through Study Completion (Approximately 5.5 Years)
  Time from First Dose of Study Treatment to First Malignancy (excluding NMSC)
Time from First Dose of Study Treatment to First Opportunistic Infection | Baseline through Study Completion (Approximately 5.5 Years)
  Time from First Dose of Study Treatment to First Opportunistic Infection
Time from First Dose of Study Treatment to First Serious Infection | Baseline through Study Completion (Approximately 5.5 Years)
  Time from First Dose of Study Treatment to First Serious Infection

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (119):
- United States (119):
  - Arizona Research Clinic PLLC, Chandler, Arizona
  - Arizona Arthritis & Rheumatology Associates, P. C., Mesa, Arizona
  - Arizona Arthritis & Rheumatology Research, Paradise Valley, Arizona
  - Sun Valley Arthritis Center, LTD, Peoria, Arizona
  - Arizona Arthritis & Rheumatology Associates, Phoenix, Arizona
  - Arthritis and Rheumatism Associates, Jonesboro, Arkansas
  - Providence St. Joseph's Medical Center, Burbank, California
  - Hope Clinical Research, Inc., Canoga Park, California
  - Medvin Clinical Research - Covina, Covina, California
  - TriWest Research Associates LLC, El Cajon, California
  - Newport Huntington Med Grp, Huntington Beach, California
  - BioSolutions Clinical Research Center, La Mesa, California
  - Valerius Medical Group and Research Center of Greater Long Beach, Los Alamitos, California
  - R. Srinivasan, M.D., Inc. dba Monterey Park Medical Center, Monterey Park, California
  - ACRC Studies, Poway, California
  - Desert Medical Advances, Rancho Mirage, California
  - Purushotham & Akther Kotha MD Inc, San Diego, California
  - East Bay Rheumatology Medical Group, Inc, San Leandro, California
  - Providence Medical Foundation, Santa Rosa, California
  - Dan La, MD Inc, Tujunga, California
  - Office: Dr Robin K Dore, Tustin, California
  - Inland Rheumatology & Osteoporosis Medical Group, Upland, California
  - Nazanin Firooz, MD Inc., West Hills, California
  - Medvin Clinical Research - Whittier, Whittier, California
  - Danbury Clinical Research, LLC, Danbury, Connecticut
  - Delaware Arthritis, Lewes, Delaware
  - Omega Research Debary, LLC, DeBary, Florida
  - Cria Center for Rheumatology, Fort Lauderdale, Florida
  - SIMED Health, Gainesville, Florida
  - GNP Research at Mark Jaffe, MD, Hollywood, Florida
  - Rheumatology Center Of Palm Beach, Pllc, Lake Worth, Florida
  - Arthritis and Rheumatology Center of South Florida, Margate, Florida
  - Miami Clinical Reserach, Miami, Florida
  - Felicidad Medical Research, Miami, Florida
  - Rheumatology Associates of Central Florida, Orlando, Florida
  - Heuer MD Research, Orlando, Florida
  - UCF Health Lake Nona Orlando, Orlando, Florida
  - IRIS Research and Development, LLC, Plantation, Florida
  - BayCare Health System Inc, St. Petersburg, Florida
  - West Broward Rheumatology Associates, Tamarac, Florida
  - Avita Clinical Research, Tampa, Florida
  - Tampa Medical Group, P.A., Tampa, Florida
  - Florida Medical Clinic LLC, Zephyrhills, Florida
  - Arthritis & Rheumatology of Georgia, Atlanta, Georgia
  - Arthritis Center of North Georgia, Gainesville, Georgia
  - St Luke's Clinic - Intermountain Orthopaedics, Boise, Idaho
  - Hinsdale Orthopaedics, Illinois Bone and Joint, Hinsdale, Illinois
  - Rockford Orthopedic Associates, Rockford, Illinois
  - Orthoillinois, Rockford, Illinois
  - Greater Chicago Specialty Physicians, LLC, Schaumburg, Illinois
  - Center of Robert Hozman, Skokie, Illinois
  - Beacon Medical Group Clinical Research, South Bend, Indiana
  - Graves-Gilbert Clinic, Bowling Green, Kentucky
  - Western KY Rheumatology PLLC, Hopkinsville, Kentucky
  - Accurate Clinical Research, Lake Charles, Louisiana
  - Arthritis and Diabetes Clinic, Inc., Monroe, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Klein and Associates MD, PA, Cumberland, Maryland
  - NECCR PrimaCare Research, Fall River, Massachusetts
  - Michigan Rheumatology Group, Grand Blanc, Michigan
  - Pandit Rheumatology PC, Okemos, Michigan
  - Jefferson City Medical Group, Jefferson City, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - West County Rheumatology, St Louis, Missouri
  - Lovelace Scientific Resources, Henderson, Nevada
  - Allied Clinical Research, Reno, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Arthritis Care Medical Center, Somerset, New Jersey
  - Atlantic Coastal Research, Toms River, New Jersey
  - Sahni Rheumatology & Therapy PC, West Long Branch, New Jersey
  - NYU Langone, New York, New York
  - Medication Management, Greensboro, North Carolina
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - Cape Fear Arthritis Care, Leland, North Carolina
  - Carolina Arthritis Associates, Wilmington, North Carolina
  - Cincinnati Arthritis Associates, Cincinnati, Ohio
  - Craig S Thompson MD LLC, Marion, Ohio
  - Paramount Medical Research, Middleburg Heights, Ohio
  - Arthritis & Rheumatology Center of Oklahoma PLLC, Oklahoma City, Oklahoma
  - Good Samaritan Hospital Corvallis, Corvallis, Oregon
  - Advanced Rheumatology and Arthritis Research Center, PC, Cranberry Township, Pennsylvania
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Pennsylvania Regional Center for Arthritis and Osteoporosis Research, Wyomissing, Pennsylvania
  - Articularis Healthcare d/b/a/ Low Country Rheumatology, PA, North Charleston, South Carolina
  - Monument Health Rapid City Hospital, Rapid City, South Dakota
  - Cumberland Rheumatology, Crossville, Tennessee
  - West Tennessee Research Institute, Jackson, Tennessee
  - Nashville Arthritis and Rheumatology, Nashville, Tennessee
  - Accent Clinical Research Professionals, LLC, Allen, Texas
  - Amarillo Center for Clinical Research, Amarillo, Texas
  - Arthritis & Osteoporosis Clinic of Brazos Valley, College Station, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - El Paso Integrated Physicians Group, P.A., an Elligo Health Research, Inc. Healthcare Enabled Research Organization, El Paso, Texas
  - UDL Clinical Research, LLC, Houston, Texas
  - Pioneer Research Solutions, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Accurate Clinical Management - Houston, Houston, Texas
  - Synergy Group US, Katy, Texas
  - Houston Rheumatology & Arthritis Specialists, Katy, Texas
  - R and H Clinical Research, Katy, Texas
  - Prime Clinical Research, Mansfield, Texas
  - Southwest Rheumatology, P.A., Mesquite, Texas
  - Advanced Clinical Research Center of Houston, Pearland, Texas
  - Clinrx Research Joseph INC., Plano, Texas
  - Violeta T. Baddour, MD, Pleasanton, Texas
  - Accurate Clinical Research, Inc., San Antonio, Texas
  - Accurate Clinical Management, Sugar Land, Texas
  - Fort Bend Clinical Research, LLC, Sugar Land, Texas
  - Mt. Olympus Medical Research, Sugar Land, Texas
  - Baylor Scott & White Health, Temple, Texas
  - North Houston Rheumatology Associates, The Woodlands, Texas
  - Dynamed Clinical Research, LP d/b/a DM Clinical Research, Tomball, Texas
  - Center for Arthritis and Rheumatic Diseases, PC, Chesapeake, Virginia
  - Spectrum Medical Inc., Danville, Virginia
  - Arthritis & Osteoporosis Center of Northern Virinia, Manassas, Virginia
  - TPMG Rheumatology/TPMG Clinical Research, Newport News, Virginia
  - Arthritis Northwest, PLLC, Spokane, Washington
  - Rheumatology & Pulmonary Clinic, Beckley, West Virginia
  - Rheumatic Disease Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Baricitinib in Participants With Rheumatoid Arthritis — https://trials.lillytrialguide.com/en-US/trial/6bOD3ngGslJ7hrvp0NfPrN